CLINICAL TRIAL: NCT04426357
Title: A Single-dose, Open-label, Parallel-group Study to Evaluate the Effect of Renal Impairment on the Pharmacokinetics of JNJ-64417184 and Its Two Minor Metabolites JNJ-68294291 and JNJ-65201526 in Adult Participants
Brief Title: A Study to Evaluate the Effect of Renal Impairment on JNJ-64417184 and Its Two Minor Metabolites JNJ-68294291 and JNJ-65201526 in Adult Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: company decision
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108800; 2019-004929-25 (EudraCT Number); 64417184RSV1008 (Other: Janssen Pharmaceutica N.V., Belgium)
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Participants with Renal impairment): JNJ-64417184 (Experimental): Participants with varying degrees of impaired renal impairment function (moderate renal impairment [optional], severe renal impairment, and end stage renal disease [ESRD] not requiring hemodialysis) will be enrolled and will receive a single oral dose of JNJ-64417184 as film coated tablet on Day 1.
  Interventions: Drug: JNJ-64417184
- Group 2 (Healthy Participants): Control Group (Active Comparator): Participants with normal renal function will be enrolled in controlled group and will receive a single oral dose of JNJ-64417184 as film coated tablet on Day 1.
  Interventions: Drug: JNJ-64417184

INTERVENTIONS:
Drug: JNJ-64417184 — Participants will receive single oral (as film coated tablet) dose of JNJ-64417184 on Day 1.

SUMMARY:
The main purpose of this study is to evaluate the pharmacokinetics of JNJ-64417184, JNJ-68294291, and JNJ-65201526 after a single oral dose of JNJ-64417184 in adult participants with various degrees of impaired renal function (moderate [optional], severe renal impairment, and end stage renal disease (ESRD) not requiring hemodialysis) compared to participants with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

* Participants with normal renal function:

must have normal renal function defined as: estimated glomerular filtration rate (eGFR) greater than or equal to (>=) 90 milliliter per minute per 1.73 meter square (mL/min/1.73 m^2 (calculated by the modification of diet in renal disease [MDRD] formula)

* Healthy on the basis of physical examination, medical and surgical history, and vital signs performed at screening. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Participants with moderate or severe renal impairment:

must meet the following additional inclusion criteria to be enrolled in the study: must be otherwise healthy except for the renal impairment and its underlying disease states and mild comorbidities and participant must be medically stable on the basis of physical examination, medical history, vital signs, 12-lead Electrocardiogram (ECG), and clinical laboratory tests performed at screening. If there are abnormalities or results outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator

* Participants with end stage renal disease (ESRD): must have a hematocrit at screening of greater than or equal to (>=) 30 percent (%)
* Must not smoke more than 10 cigarettes or 2 cigars or 2 pipes per day from within 3 months prior to screening until the end of the study

Exclusion Criteria:

* History of any illness (unrelated to renal impairment or its underlying disease, as appropriate) that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant. This may include but is not limited to history of relevant drug or food allergies, history of cardiovascular or central nervous system disease, history or presence of clinically significant pathology, chronic skin disease, or history of mental disease
* Known allergies, hypersensitivity, or intolerance to JNJ-64417184 or any of its excipients
* Past history of clinically significant cardiac arrhythmias (example, extrasystole, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (example, hypokalemia, family history of long QT Syndrome)
* Any evidence of clinically significant heart block or bundle branch block at screening
* Current human immunodeficiency virus type 1 (HIV-1) or HIV-2 infection (confirmed by antibodies) at screening
* History of hepatitis A, B, or C infection, or current hepatitis A infection (confirmed by hepatitis A antibody immunoglobulin M [IgM]), or hepatitis B virus (HBV) infection (confirmed by hepatitis B surface antigen), or hepatitis C virus (HCV) infection (confirmed by HCV antibody) at screening

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Analyte Concentration (Cmax) of JNJ-64417184and its Metabolites (JNJ-68294291 and JNJ-65201526) | Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, 120 and 216 hours post dose
  Cmax is defined as maximum observed plasma analyte concentration of JNJ-64417184 and its metabolites (JNJ-68294291 and JNJ-65201526).
Area under the Plasma Analyte Concentration Time Curve from Time 0 to Time of the Last Measurable Concentration [AUC (0-Last)] of JNJ-64417184 and its Metabolites (JNJ-68294291 and JNJ-65201526) | Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, 120 and 216 hours post dose
  AUC (0-Last) is defined as area under the plasma analyte concentration time curve from time 0 to time of the last measurable (non-below quantification limit [BQL]) concentration of JNJ-64417184 and its metabolites (JNJ-68294291 and JNJ-65201526).
Area Under the Plasma Analyte Concentration Time Curve from Time 0 to Infinite Time [AUC (0-Infinity)] of JNJ-64417184 and its Metabolites (JNJ-68294291 and JNJ-65201526) | Predose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72, 96, 120 and 216 hours post dose
  AUC (0-infinity) is defined as area under the plasma analyte concentration time curve from time 0 to infinite time, calculated as AUC (last) plus C(last)/(lambda)z, where C (last) is the last observed measurable (non-BQL) plasma analyte concentration; extrapolations of more than 20 percent (%) of the total AUC (that is, percent AUC (infinity), extrapolations greater than [>] 20%) are reported as approximations of JNJ-64417184 and its metabolites (JNJ-68294291 and JNJ-65201526).

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to Day 11
  An AE is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium Clinical Trial, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (2):
- Germany (2):
  - CRS Clinical Research Services Kiel GmbH, Kiel
  - APEX GmbH, München

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency